CLINICAL TRIAL: NCT04303260
Title: Special Physical Exercises as a Therapeutic Intervention for Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Shmuel Kivity, MD, Director of Clinical Research and Development Department, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0277-18-TLV
Record Dates: First submitted 2019-07-01; First posted 2020-03-11 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm (Active Comparator): Patients in the interventional arm will be asked to complete 3 different videos repeatedly, as many days a week as possible. This repetition is to be maintained even if a patient missed one day of training.
  The interventional exercise regimen will include specific exercises postulated to increase blood flow to the intestine and colon and thereby promote normal peristaltic s and decrease inflammation.
  Interventions: Behavioral: Physical exercises
- controled arm (Placebo Comparator): Patients in the controled arm will also be asked to practice generally recommended exercises in 3 different videos repeatedly, as many sets as possible..
  The control arm will practice generally recommended exercises, without particular attention to the abdomen.
  Interventions: Behavioral: Physical exercises

INTERVENTIONS:
Behavioral: Physical exercises — The interventional exercise regimen will include specific exercises postulated to increase blood flow to the intestine and colon and thereby promote normal peristaltic s and decrease inflammation.

SUMMARY:
The investigator is hypothesize that physical activity can have positive effects on health, general well-being , sleep quality and stress in Inflammatory Bowel Disease patients.

DETAILED DESCRIPTION:
A randomized-controlled-double blinded pilot study. 50 Inflammatory Bowel Disease patients, suffering from mild disease will be randomized to undergo either a set of specific physical exercises for Inflammatory Bowel Disease or a control set of unrelated exercises.

Patients will be randomized to either interventional or control groups by a computer automatized randomization program. Patients will be sent an email with the link to an internet site where they will be able to watch the exercise program.

The interventional exercise regimen will include specific exercises postulated to increase blood flow to the intestine and colon and thereby promote normal peristaltic and decrease inflammation. The control arm will practice generally recommended exercises, without particular attention to the abdomen.

Videos of sets of exercise will be available online which patients will be able to watch and follow from their home computer. The exercise regimens (both interventional and controls) will be sequenced and performed by a trained and experienced instructor, which will provide these to the PI. Each video will include explicit instructions and examples for each of the exercises. Patients will be asked to watch the videos and preform the exercises individually every day. Patients in the interventional arm will be asked to complete 3 different videos repeatedly, as many days a week sets as possible. This repetition is to be maintained even if a patient missed one day of training to perform sets of 15 minutes/ day, 6 times a week.; Compliance will be documented by patients through emails to the study coordinator. Patients in the controled arm will also be asked to practice generally recommended exercises in 3 different videos repeatedly, as many sets as possible.

Patients will answer questionnaires once every two weeks(week 0, 2, 4). Patients will answer QOL(quality of life), PROMs(Patient Reported Outcome Measures),disease activity , Sleep questionnaire and Morningness eveningness questionnaire. Also, before and after the intervention (week 0 and week 4) patients will visit the clinic for anthropometric measurements and to give serum, stool and urine sample which will be analyzed for inflammatory markers, microbial composition and function.

ELIGIBILITY:
Inclusion Criteria:

1. 18 < age < 60
2. Clinically stable patients, constant medicinal regimen throughout the study period. Refractory to mesalamine at least 6 weeks, or steroids at least 2 week, or immunomodulator at least 12 weeks or biologics at least 12 weeks therapy, medical cannabis at least 2 weeks before the study.
3. CD patients will be included if their symptoms score 5≤ between ≤15 on the Harvey-Bradshaw index (HBI) score
4. UC patients will be included if their symptoms score 3≤between≤9 on the Simple Clinical Colitis Activity Index (SCCAI)

Exclusion Criteria:

1. Inability to commit for performing at least 15 minutes of exercise, 6 times a week
2. Lack of availability or capability to use a computer/ internet.
3. Any proven current infection such as Clostridium difficile infection, positive stool culture, or parasites.
4. Inability to sign informed consent and complete study protocol
5. Pregnancy
6. Subjects with chronic conditions such as cancer, organ transplant subjects, advanced kidney or liver disease, systemic inflammatory conditions other than IBD.
7. Patients with ileostomy, pouch or short bowel

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Clinical response assessed by a change in HBI | After 4 weeks
  Doctor evaluation -The Harvey-Bradshaw index activity index
  Harvey Bradshaw Index (based on the day before):
  General well-being:
  * very well =0
  * slightly below par =1
  * poor =2
  * very poor =3
  * terrible =4
  Abdominal pain:
  * none =0
  * mild =1
  * moderate =2
  * severe =3
  Abdominal mass:
  * none =0
  * dubious =1
  * definite =2
  * definite and tender =3
  Number of liquid stools per day:
  Complications:
  * none =0
  * arthralgia =1
  * uveitis =1
  * erythema nodosum =1
  * aphthous ulcers =1
  * pyoderma gangrenosum =1
  * anal fissure =1
  * new fistula =1
  * abscess =1
  SCORE:
  <5 Remission 5-7 Mild activity 8-16 Moderate activity >16 Sever activity
Clinical response as assessed by a change in SCCAI | After 4 weeks
  Doctor evaluation- Simple Clinical Colitis Activity Index
  Bowel frequency (day):
  * 0-3 / day (0)
  * 4-6 / day (1)
  * 7-9 / day (2)
  * >9 / day (3)
  Bowel frequency (night):
  * 0 / night (0)
  * 1-3 / night (1)
  * 4-6 / night (2)
  General well being:
  * very well (0)
  * slightly below par (1)
  * poor (2)
  * very poor (3)
  * terrible (4)
  Urgency of defecation:
  * none (0)
  * Hurry (1)
  * Immediately (toilet nearby) (2)
  * Incontinence (3)
  Blood in stool:
  * None (0)
  * Trace (1)
  * Occasionally (<50% of defecations) (2)
  * Usually (>50% of defecations) (3)
  SCCAI Score:
  (add scores of questions 1 to 5) Remission<3 Mild Disease 3-5 Moderate Disease 6-9 Severe Disease ≥10
Clinical response as assessed by a change in PROMIS questionnaire | After 4 weeks
  PROMIS (Patient-Reported Outcomes Measurement Information System)
Clinical response as assessed by a change in QOL questionnaire | After 4 weeks
  Quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nitsan Maharshak, MD, Principal Investigator — Tel Aviv Medical Center- Head of Inflammatory Bowel Disease Center
Locations (1):
- Dep. of Gastroenterology, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No